CLINICAL TRIAL: NCT07214662
Title: A Phase Ia/Ib Dose-Escalation and Expansion Study Evaluating the Safety, Pharmacokinetics, and Activity of GDC-0587 as a Monotherapy and in Combination With Giredestrant in Patients With Locally Advanced Or Metastatic ER-Positive, HER2-Negative Breast Cancer Who Have Previously Progressed During or After CDK4/6 Inhibitor Therapy
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of GDC-0587 as a Monotherapy and in Combination With Giredestrant in Participants With Locally Advanced or Metastatic Estrogen Receptor-Positive and Human Epidermal Growth Factor Receptor 2-Negative (ER+/HER2-) Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO46057
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase Ia: GDC-0587 Monotherapy (Experimental): Participants will receive GDC-0587 orally.
  Interventions: Drug: GDC-0587
- Phase Ib: GDC-0587 + Giredestrant Cohort (Experimental): Participants will receive GDC-0587 and Giredestrant orally.
  Interventions: Drug: GDC-0587; Drug: Giredestrant
- Phase Ib: GDC-0587 + Giredestrant Food-Effect and PPI-Effect Cohort (Experimental): Participants will receive GDC-0587 and Giredestrant orally and also receive omeprazole for evaluating the effects of a proton pump inhibitor (PPI) and food on GDC-0587.
  Interventions: Drug: GDC-0587; Drug: Giredestrant; Drug: Omeprazole

INTERVENTIONS:
Drug: GDC-0587 — Participants will receive GDC-0587 orally as per the schedule in the protocol.
  Other Names: RO7840736; RGT-587
Drug: Giredestrant — Participants will receive Giredestrant orally as per the schedule in the protocol.
  Other Names: GDC-9545; RO7197597; RG6171
  Arms: Phase Ib: GDC-0587 + Giredestrant Cohort; Phase Ib: GDC-0587 + Giredestrant Food-Effect and PPI-Effect Cohort
Drug: Omeprazole — Participants will receive Omeprazole orally as per the schedule in the protocol.
  Arms: Phase Ib: GDC-0587 + Giredestrant Food-Effect and PPI-Effect Cohort

SUMMARY:
This is a first-in-human, Phase Ia/Ib, dose-escalation and expansion study evaluating the safety, pharmacokinetics, and activity of GDC-0587 (cyclin-dependent kinase-4 [CDK4] inhibitor) as a monotherapy and in combination with giredestrant in participants with locally advanced or metastatic estrogen receptor-positive and human epidermal growth factor receptor 2-negative (ER+/HER2-) breast cancer who have previously progressed during or after CDK 4/6 inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to adhere to the contraception requirements
* For females of childbearing potential ≤60 years of age and males: treatment with luteinizing hormone-releasing hormone (LHRH) agonist therapy beginning at least 2 weeks prior to Cycle 1, Day 1 and agreement to continue LHRH agonist therapy for the duration of the study
* Histologically or cytologically confirmed adenocarcinoma of the breast that is locally advanced or metastatic
* Previously documented ER+ and HER2- tumor according to American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) or European Society of Medical Oncology (ESMO) guidelines or any national guidelines with criteria conforming to ASCO/CAP or ESMO guidelines
* Disease progression during or following treatment with an approved CDK 4/6 inhibitor, with or without endocrine therapy, in the locally advanced or metastatic setting
* Measurable, or non-measurable but evaluable, disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥6 months
* Creatinine clearance ≥60 milliliter per minute (mL/min) (calculated through use of the Cockcroft-Gault formula)

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant during the study
* Advanced, symptomatic, visceral spread that is at risk of life-threatening complications in the short term appropriate for treatment with cytotoxic chemotherapy at time of entry into the study, as per national or local treatment guidelines
* Five or more prior lines of systemic therapy in the locally advanced or metastatic setting
* Treatment with anti-cancer therapies, including investigational therapies, within 28 days or 5 drug elimination half-lives, whichever is shorter, prior to initiation of study drug
* Treatment with an approved oral endocrine therapy within 7 days prior to initiation of study drug or treatment with fulvestrant or an approved/investigational CDK inhibitor within 21 days prior to initiation of study drug
* History of Grade ≥3 adverse event attributed to prior CDK inhibitor therapy that resulted in permanent discontinuation of prior CDK inhibitor therapy
* Poor peripheral venous access
* Malabsorption condition or other gastrointestinal (GI) conditions/surgeries that the investigator assesses may significantly interfere with enteral absorption
* Major surgical procedure within 28 days prior to initiation of study drug
* Untreated, active CNS metastases
* Infection requiring systemic (i.e., oral, IV, or intramuscular) antibiotics, chronic infection requiring treatment within 1 year prior to screening, or any evidence of current infection
* History of malignancy within 3 years prior to screening, except for cancer under investigation in this study
* Known history of a clinically significant abnormal ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | From Baseline to 30 days after final dose of study treatment (Up to approximately to 18 months)
  Measured by reporting the incidence and severity using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 grading scale.
Percentage of Participants with Dose-limiting Toxicity (DLTs) | Phase 1a: Days 1-28 of Cycle 1; Phase 1b: Days 1-28 of Cycle 1 (Each cycle is 28 days)

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response Rate (ORR) of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Up to approximately to 18 months
Plasma Concentration of GDC-0587 as a Monotherapy and in Combination With Giredestrant | Phase 1a: Cycle 1 (Day 1, 2 15, 16), Cycle 2, 3, 5, 7, 9, 11 (Day 1); Phase 1b: Cycle 1 (Day 1, 2 15, 16), Cycle 2, 3, 5, 7, 9, 11 (Day 1) (Each cycle is 28 days)
Plasma Concentration of GDC-0587 with Giredestrant Under Fasted and Fed Conditions | Part 1b: Cycle 1 (Day 1, 2, 4), Cycle 2, 3, 5, 7, 9 and 11 (Day 1) (Each cycle is 28 days)
Plasma Concentration of GDC-0587 with Giredestrant Following Multiple-dose Administration, Either Alone or in Combination With Omeprazole | Part 1b: Cycle 1 (Day 11, 12, 20 and 21) (Each cycle is 28 days)
Recommended Phase II Dose (RP2D) of GDC-0587 | Up to approximately to 18 months
Recommended Phase II Dose (RP2D) of GDC-0587 in Combination with Giredestrant | Up to approximately to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (2):
- United States (2):
  - START - Midwest - EDOS, Grand Rapids, Michigan
  - START - San Antonio - EDOS, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No